CLINICAL TRIAL: NCT02613845
Title: Predictors for Postoperative Delirium After Cardiac Surgery in Adults: a One-year, Single Center, Observational Cohort Study
Acronym: PODCAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Nicolai Goettel, MD, DESA, EDIC, University Hospital, Basel, Switzerland
Other Study IDs: PODCAS
Record Dates: First submitted 2015-11-17; First posted 2015-11-25 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; Cardiac surgery; Cardiopulmonary bypass; Risk factor
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery: Study subjects are all patients who underwent cardiac surgery with cardiopulmonary bypass at the University Hospital Basel during the year 2013.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
The Diagnostic and Statistical Manual of Mental Disorders, 5th ed. (DSM-5) describes delirium as a "disturbance in attention (i.e., reduced ability to direct, focus, sustain, and shift attention) and awareness (reduced orientation to the environment)". In addition, a "disturbance in cognition (e.g., memory deficit, disorientation, language, visuospatial ability, or perception)" occurs.

Postoperative delirium (POD) usually develops in connection with a surgical procedure within the first five days after an intervention. Roughly 10-70% of all surgical patients above the age of 65 years are affected.

POD places not only a burden to the patient and their families by increasing functional and cognitive damages, and increasing mortality, it also has a high impact on the health care resource utilization. A patient with POD often requires more intensive care, has a longer length of hospital stay, more complications, and often requires long-term care after being discharged from the hospital. All these aspects show the need for prevention of POD.

There are various preoperative risk factors that influence the development of POD. Broad research has been done on this topic and shown that advanced age, cognitive impairment, depression and other psychopathologic symptoms, intake of psychotropic substances, sensory impairment like decrease in visual or auditory perception, impairment in daily life activities, dehydration, malnutrition, metabolic dysfunctions, urinary catheters, severity of disease and different comorbidities, such as chronic cardiac insufficiency, atrial fibrillation, or previous history of stroke or infections may favor the occurrence of POD.

The incidence of POD is among the highest in cardiac surgery. The study was designed to assess predictors for POD after cardiac surgery. Study hypothesis is that some patient variables, scores and biomarkers are not only predictive of the incidence of POD but also of the severity of delirium-associated symptoms and duration of POD after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

All patients who underwent cardiac surgery with cardiopulmonary bypass at University Hospital Basel in 2013 were included.

Exclusion Criteria:

* Patients who died during the operation.
* Patients who lack the primary outcome measure.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects are all patients who underwent cardiac surgery at the University Hospital Basel during the year 2013. Patients are identified by screening of the list of operative procedures of this year, made available by the Department of Cardiac Surgery at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 656 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | Baseline value on postoperative day 1 and postoperative day 2 until discharge from the intensive care unit
  Postoperative delirium diagnosed by the Intensive Care Delirium Screening Checklist (ICDSC)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No